CLINICAL TRIAL: NCT04707456
Title: A Comparative Study of Learning Curve Between Two Different Levels of Proficiency for First Trimester Fetal Anomaly Scan Using ISUOG Guidelines
Brief Title: Comparative Study of Learning Curve for First Trimester Fetal Anomaly Scan
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Saranthorn Sripilaipong, Doctor, Mahidol University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: COA. MURA2020/303
Record Dates: First submitted 2021-01-11; First posted 2021-01-13 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: First Trimester Pregnancy
Keywords: First trimester ultrasound scan; Learning curve; ISUOG practice guidelines

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MFM staff-level operator (No Intervention)
- MFM fellowship trainee-level operator (Other)
  Interventions: Other: Training operator

INTERVENTIONS:
Other: Training operator — After recruitment, the participants were divided into two groups to perform first-trimester ultrasound scan by two different levels of proficiency.
  First group : operator has experience more than 3 years in NT scan and second trimester ultrasound scan Second group : operator has experience less than 3 years in NT scan and second trimester ultrasound scan
  Arms: MFM fellowship trainee-level operator

SUMMARY:
Ultrasound scans during first trimester are more difficult than routine mid-trimester ultrasound scans. Practice guidelines for first trimester fetal ultrasound scans have been provided by the International Society of Ultrasound in Obstetrics and Gynecology (ISUOG) since 2013. Using this guidelines, different levels of proficiency operators might have equal ability to complete first trimester ultrasound scans.

DETAILED DESCRIPTION:
Nowadays, high-resolution transabdominal ultrasounds are widely used, and ultrasound scans for fetal structural abnormalities at the first trimester are indeed possible. First trimester ultrasound scans are important and essential for detecting fetal structural anomalies, and they help provide optimized early antenatal management. However, ultrasound scans, during this period, are more difficult than routine mid-trimester ultrasound scans, as fetal organs are small and experienced operators are needed to use the transducer to obtain informative pictures. Practice guidelines for first trimester fetal ultrasound scans have been provided by the International Society of Ultrasound in Obstetrics and Gynecology (ISUOG) since 2013. Since then, the percentage of complete scans and the high detection rate of fetal structural abnormalities during first trimester ultrasound scans have been reported. From our perspective, ultrasound operators who have different experiences in mid-trimester ultrasound scanning might have equal ability to complete first trimester ultrasound scans using the ISUOG guidelines. The objective of this study is to compare the rate of completed scans regarding fetal structures at the first trimester ultrasound scan between two different levels of proficiency operators.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Maternal age ≥ 18 years
* Gestational age between 11-13 + 6 weeks by last menstrual date or ultrasound report if uncertain date

Exclusion Criteria:

* Multifetal gestation
* Miscarriage before first trimester ultrasound
* Loss to follow up at mid-trimester ultrasound scan
* Loss to follow up after birth

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2020-06-11 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Percent of completed scans of fetal structural abnormality between two different levels of proficiency operators | 3 months
  To compare the percentage of completed scans of each organ during the first trimester scan between two different levels of proficiency

SECONDARY OUTCOMES:
Screening time for first trimester ultrasound scans between two different levels of proficiency operators | 3 months
  To compare screening time for first trimester ultrasound scans between two different levels of proficiency operators
Learning curve of first trimester ultrasound scans between two different levels of proficiency operators | 3 months
  To compare the learning curve between two different levels of proficiency operators
Detection rate of fetal structural abnormality in first trimester ultrasound scans between two different levels of proficiency operators | 9 months
  To compare the detection rate of fetal structural abnormality between two different levels of proficiency operators

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology, Faculty of Medicine Ramathibodi hospital, Mahidol university, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Centers for Disease Control and Prevention (CDC). Update on overall prevalence of major birth defects--Atlanta, Georgia, 1978-2005. MMWR Morb Mortal Wkly Rep. 2008 Jan 11;57(1):1-5. PMID 18185492
- [Background] Pangkanon S, Sawasdivorn S, Kuptanon C, Chotigeat U, Vandepitte W. Establishing of National Birth Defects Registry in Thailand. J Med Assoc Thai. 2014 Jun;97 Suppl 6:S182-8. PMID 25391192
- [Background] Karim JN, Roberts NW, Salomon LJ, Papageorghiou AT. Systematic review of first-trimester ultrasound screening for detection of fetal structural anomalies and factors that affect screening performance. Ultrasound Obstet Gynecol. 2017 Oct;50(4):429-441. doi: 10.1002/uog.17246. Epub 2017 Sep 7. PMID 27546497
- [Background] Taipale P, Ammala M, Salonen R, Hiilesmaa V. Learning curve in ultrasonographic screening for selected fetal structural anomalies in early pregnancy. Obstet Gynecol. 2003 Feb;101(2):273-8. doi: 10.1016/s0029-7844(02)02590-5. PMID 12576250
- [Background] Salomon LJ, Alfirevic Z, Bilardo CM, Chalouhi GE, Ghi T, Kagan KO, Lau TK, Papageorghiou AT, Raine-Fenning NJ, Stirnemann J, Suresh S, Tabor A, Timor-Tritsch IE, Toi A, Yeo G. ISUOG practice guidelines: performance of first-trimester fetal ultrasound scan. Ultrasound Obstet Gynecol. 2013 Jan;41(1):102-13. doi: 10.1002/uog.12342. No abstract available. PMID 23280739
- [Background] Srisupundit K, Tongsong T, Sirichotiyakul S, Chanprapaph P. Fetal structural anomaly screening at 11-14 weeks of gestation at Maharaj Nakorn Chiang Mai Hospital. J Med Assoc Thai. 2006 May;89(5):588-93. PMID 16756041
- [Background] Petousis S, Sotiriadis A, Margioula-Siarkou C, Tsakiridis I, Christidis P, Kyriakakis M, Mamopoulos A, Athanasiadis A, Dagklis T. Detection of structural abnormalities in fetuses with normal karyotype at 11-13 weeks using the anatomic examination protocol of the International Society of Ultrasound in Obstetrics and Gynecology (ISUOG). J Matern Fetal Neonatal Med. 2020 Aug;33(15):2581-2587. doi: 10.1080/14767058.2018.1555807. Epub 2019 Jan 7. PMID 30612473
- [Background] Nicolaides KH. Nuchal translucency and other first-trimester sonographic markers of chromosomal abnormalities. Am J Obstet Gynecol. 2004 Jul;191(1):45-67. doi: 10.1016/j.ajog.2004.03.090. PMID 15295343
- [Background] Salvesen K, Lees C, Abramowicz J, Brezinka C, Ter Haar G, Marsal K; Board of International Society of Ultrasound in Obstetrics and Gynecology (ISUOG). ISUOG statement on the safe use of Doppler in the 11 to 13 +6-week fetal ultrasound examination. Ultrasound Obstet Gynecol. 2011 Jun;37(6):628. doi: 10.1002/uog.9026. No abstract available. PMID 21618313